CLINICAL TRIAL: NCT03155919
Title: Effects of Taurine and Chocolate Milk Supplementation in Body Composition, Athletic Performance and Oxidative Stress in Triathletes.
Brief Title: Taurine Supplementation and Triathletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ellen Cristini de Freitas, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AN FCFAR UNESP
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Athletic Proteinuria
Keywords: taurine; triathletes; oxidative stress; chocolate milk

STUDY DESIGN:
Intervention Model Description: A double-blind, crossover, 2-week washout study will be conducted with 20 male triathletes, aged 30 to 45 years, which will be offered during eight weeks capsules containing three grams of taurine or placebo and 400 ml of chocolate milk ready to drink.
Who Masked: Participant, Investigator
Masking Description: The taurine and placebo powder were offered in capsules identified by Taurine A and Taurine B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAUchoc (Experimental): Treatment composed by taurine powder and chocolate milk
  Interventions: Dietary Supplement: TAUchoc
- PLAchoc (Placebo Comparator): Treatment composed by placebo (starch powder) and chocolate milk
  Interventions: Dietary Supplement: PLAchoc

INTERVENTIONS:
Dietary Supplement: TAUchoc — The supplements were offered during eight weeks in capsules containing three grams of taurine powder and 400 ml of chocolate milk ready to drink.
  Arms: TAUchoc
Dietary Supplement: PLAchoc — The supplements were offered during eight weeks in capsules containing three grams of placebo (starch powder) and 400 ml of chocolate milk ready to drink.
  Arms: PLAchoc

SUMMARY:
Taurine is a nitrogenous compound, naturally present in heart, leukocytes, retina, central nervous system, especially in muscles. It has several beneficial physiological effects like antioxidant action, and could increase muscle force contraction and insulin sensibility. Triathlon is a sport of medium to high intensity, that can causes an increase in the rate of oxygen consumption during intense exercise and consequently increases free radicals production and oxidative stress, which may compromise an athlete's performance. Due to the weekly intense training, triathletes need nutritional care ranging from calories and nutrients adequacy to the use of specific nutrients that can help to maintain health. Thus, it is believed that the use of taurine associated with chocolate milk after exercise can promote general metabolic insulin action in order to favor carbohydrates metabolism regulation, assist muscle recover and prevent oxidative damage and thus promote triathletes performance and muscle mass gain. Thus, the aim of this project is to evaluate the effects of taurine and chocolate milk supplementation in body composition, athletic performance and oxidative stress in triathletes.

DETAILED DESCRIPTION:
BACKGROUND: Taurine is a nitrogenous compound, naturally present in heart, leukocytes, retina, central nervous system, especially in muscles. It has several beneficial physiological effects like antioxidant action, and could increase muscle force contraction and insulin sensibility. Triathlon is a sport of medium to high intensity, that can causes an increase in the rate of oxygen consumption during intense exercise and consequently increases free radicals production and oxidative stress, which may compromise an athlete's performance. Due to the weekly intense training, triathletes need nutritional care ranging from calories and nutrients adequacy to the use of specific nutrients that can help to maintain health. Thus, it is believed that the use of taurine associated with chocolate milk after exercise can promote general metabolic insulin action in order to favor carbohydrates metabolism regulation, assist muscle recover and prevent oxidative damage and thus promote triathletes performance and muscle mass gain.

OBJECTIVE: Evaluate the effects of taurine and chocolate milk supplementation in body composition, athletic performance and oxidative stress in triathletes MÉTHODS: A double-blind, crossover, 2-week washout study will be conducted with 20 male triathletes, aged 30 to 45 years, which will be offered during eight weeks capsules containing three grams of taurine or placebo and 400 ml of chocolate milk ready to drink. In order to assess the effects of supplementation, concentrations of serum and urinary taurine, lactate, insulin, insulin sensitivity (HOMA-IR), markers of protein metabolism (urinary nitrogen, creatinine and urea) and oxidative stress markers (MDA, GSH and vitamin E) will be quantified. Body composition will be measured by the method of deuterium labeled water. The evaluations will occur in four stages: 1o - before starting the training season; 2o - after 8 weeks of training; 3o- before starting the second training season; and 4o- after 8 weeks of training and supplementation completion. Data will be organized according to the study groups on average and standard deviation with application of analysis of variance test for verifying significant differences

ELIGIBILITY:
Inclusion Criteria:

* male, long distance triathletes, who competed in semiprofessional triathlons. Their training was focused on the Brazilian Ironman Championships.

Exclusion Criteria:

* Participants were excluded if they had experienced muscle injury in the past six months and/or were currently taking chronic or daily doses of anti-inflammatory medication or nutritional supplements.
* Participants who had a history of cardiovascular diseases.

Ages: 30 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline taurine plasma levels at 8 weeks | 8 weeks
  Plasma taurine was determined by high-performance liquid chromatography (Shimadzu, model LC 10AD). Taurine 99 % was used as standard (Sigma-Aldrich, St. Louis, MO, USA) following the method of Deyl et al (1986).

SECONDARY OUTCOMES:
Evaluation of the effects of taurine and chocolate milk supplementation on protein metabolism markers of triathletes. | Pre and Post the 8 weeks of treatment
  Determination of blood creatinine and urea by Labtest Kit, and quantification of urinary excretion of nitrogen according to the method proposed by Grimble et al. (1988).
Evaluation of the effects of taurine and chocolate milk supplementation on triathletes aerobic performance | Pre and Post the 8 weeks of treatment
  All subjects performed a maximal incremental running test with 1% gradient on a treadmill (Super ATL, Inbramed, Brazil) in a controlled environment. The test began at 8 km·h-1 and speed was increased by 1 km·h-1 every three minutes until volitional exhaustion.
Evaluation of the effects of taurine and chocolate milk supplementation on oxidative stress of triathletes. | Pre and Post the 8 weeks of treatment
  Oxidative stress markers indicative of lipid peroxidation determined: reduced glutathione (GSH) according to the method of Sedlak and Lindsay (1968) and malondialdehyde (MDA) using the method proposed by Gerard-Monnier et al. (Gerard-Monnier et al. 1998).

CONTACTS AND LOCATIONS:
Locations (1):
- Flavia Giolo de Carvalho, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
IPD won´t be available